CLINICAL TRIAL: NCT00271609
Title: A Phase II Trial of Bevacizumab for Patients With Recurrent High-Grade Gliomas
Brief Title: Bevacizumab for Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Teri Kreisl, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060064; 06-C-0064; NCT00290797 (obsolete NCT alias)
Record Dates: First submitted 2005-12-31; First posted 2006-01-02 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent High-Grade Gliomas; Malignant Gliomas
Keywords: AVASTIN; Recurrence; Chemotherapy; Anti-Angiogenesis; Radiotherapy; Brain Tumor; Malignant Glioma
MeSH Terms: conditions — Glioma; Recurrence; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anaplastic Glioma (AG) (Other): Anaplastic astrocytoma Anaplastic oligodendroglioma Anaplastic mixed oligoastrocytoma Malignant astrocytoma (not otherwise specified) 10 mg/kg intravenously over 90 minutes every 2 weeks on a 28 day cycle. First dose is given over 90 minutes and subsequent doses are given over 30 minutes.
  Interventions: Drug: Bevacizumab
- Glioblastoma Multiforme (GBM) (Other): Glioblastoma multiforme Gliosarcoma 10 mg/kg intravenously over 90 minutes every 2 weeks on a 28 day cycle. First dose is given over 90 minutes and subsequent doses are given over 30 minutes.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg intravenously over 90 minutes every 2 weeks on a 28 day cycle. First dose is given over 90 minutes and subsequent doses are given over 30 minutes.
  Other Names: rhuMAb VEGF

SUMMARY:
Background:

Bevacizumab is a genetically engineered antibody that blocks the growth of new blood vessels in tumors. Inhibiting the formation of these blood vessels may slow or stop disease progression by diminishing the supply of life-sustaining nutrients and oxygen the blood delivers to the tumor.

Bevacizumab is approved for treating colorectal cancer and has shown activity against brain tumor cells in laboratory and animal tests.

Objectives:

To examine the safety and side effects of bevacizumab in patients with recurrent brain tumors.

To determine the anti-tumor activity of bevacizumab in patients with recurrent brain tumors.

Eligibility:

Patients 18 years of age and older with a brain tumor that continues to grow after receiving standard treatments.

Design:

Patients complete the following procedures during the study:

* Infusions of bevacizumab through a vein once every 2 weeks in 4-week treatment cycles.
* Positron emission tomography (PET) scan before the first dose of bevacizumab, at the end of the first treatment cycle, and as needed after that.
* Magnetic resonance imaging (MRI) scan before the first dose of bevacizumab, within 48-96 hours after the first dose of bevacizumab in the first treatment cycle, and then every 4 weeks. One tube of blood for research is collected at the time of each MRI scan to look at specific cells.
* Physical and neurological examinations every 2 weeks for the first treatment cycle and then every 4 weeks.
* Quality-of-life questionnaires every 4 weeks.

DETAILED DESCRIPTION:
Background

* In vivo experiments have documented the ability of anti-vascular endothelial growth factor (VEGF) antibodies like bevacizumab to inhibit tumor growth in various preclinical tumor models, including gliomas.
* Given the pronounced neovasculature associated with over-expression of VEGF in malignant gliomas, and abundant published data demonstrating the dependence of glioma growth on the maintenance and proliferation of this neovasculature, bevacizumab represents a potentially promising new therapeutic approach to these otherwise refractory tumors.

Objective

* To establish data regarding the anti-tumor activity of bevacizumab in patients with recurrent high-grade gliomas as determined by progression-free-survival.
* To obtain information regarding the safety of bevacizumab administered to patients with recurrent high-grade gliomas.

Eligibility

* Adult patients with histologically proven intracranial malignant glioma
* Patients must have evidence for tumor progression by magnetic resonance imaging (MRI) scan
* Patients must have progressed after radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry

Design

* Patients will be treated with bevacizumab by intravenous injection at a dose of 10mg/kg every two weeks on a 4-week cycle.
* Prior to the first dose of bevacizumab and at the completion of the first 4-weeks of treatment, patients will undergo a fludeoxyglucose 18F -positron emission tomography (FDG-PET) scan (in cycle one only and then as needed) and a MRI perfusion scan.
* Peripheral blood circulating endothelial progenitor cells will be collected at the time of each MRI-perfusion scan. Additionally, patients will undergo a MRI perfusion scan within 48-96 hours of their first dose of bevacizumab (in cycle one only).
* For patients who are clinically/neurologically stable and with stable or responding radiographic disease at the end of each treatment cycle, treatment will continue with bevacizumab every 2 weeks, repeating MRI-perfusion scans at the conclusion (e.g. prior to another administration of bevacizumab) of each 4 week cycle.

A total of 88 patients will be enrolled on this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically proven intracranial malignant glioma will be eligible for this protocol.
* Malignant glioma include glioblastoma multiforme (GBM),
* gliosarcoma,
* anaplastic astrocytoma (AA),
* anaplastic oligodendroglioma (AO),
* anaplastic mixed oligoastrocytoma (AMO),
* or malignant astrocytoma NOS (not otherwise specified).
* Patients must have evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* This scan should be performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days.
* If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required.
* The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:
* They have recovered from the effects of surgery.
* Residual disease following resection of recurrent tumor is not mandated for eligibility into the study.
* To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:
* no later than 96 hours in the immediate post-operative period or
* at least 4 weeks post-operatively, and
* within 14 days of registration, and
* on a steroid dosage that has been stable for at least 5 days.
* If the 96 hour scan is more than 21 days before registration, the scan needs to be repeated.
* If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
* Patients must have progressed after radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be greater than or equal to 18 years old,
* and with a life expectancy greater than 8 weeks.
* Patients must have a Karnofsky performance status of greater than or equal to 60.
* Patients must have recovered from the toxic effects of prior therapy:
* 2 weeks from any investigational agent,
* 4 weeks from prior cytotoxic therapy,
* two weeks from vincristine,
* 6 weeks from nitrosoureas,
* 3 weeks from procarbazine administration,
* and 1 week for non-cytotoxic agents, e.g., interferon,
* tamoxifen,
* thalidomide,
* cis-retinoic acid, etc. (radiosensitizer does not count).
* Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
* Patients must have adequate bone marrow function (white blood count (WBC) -greater than or equal to 3,000/microliters,
* absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3,
* platelet count of greater than or equal to 100,000/mm^3,
* and hemoglobin greater than or equal to 10 gm/dl),
* adequate liver function (serum glutamic oxaloacetic transaminase (SGOT) and -bilirubin less than 2 times upper limit of normal (ULN)),
* and adequate renal function (creatinine less than 1.5 mg/dL and/or creatinine -clearance greater than or equal to 60 cc/min) before starting therapy.
* These tests must be performed within 14 days prior to registration. -Eligibility level for hemoglobin may be reached by transfusion.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects.
* Males and females will be recruited with no preference to gender.
* No exclusion to this study will be based on race.
* Minorities will actively be recruited to participate.
* Urine protein should be screened by dipstick or urine analysis for Urine Protein Creatinine (UPC) ratio.
* For proteinuria greater than or equal to 1+ or urine protein:
* creatinine UPC ratio greater than 1.0,
* 24-hour urine protein should be obtained and the level should be less than 1000 mg for patient enrollment.
* Patients must practice adequate contraception

EXCLUSION CRITERIA:

* Patients who, in the view of the treating physician,
* have significant active cardiac,
* hepatic,
* renal,
* or psychiatric diseases are ineligible.
* No concurrent use of other standard chemotherapeutics or investigative agents.
* Patients known to have a malignancy that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except non-melanoma skin cancer or carcinoma in-situ in the cervix).
* Patients who have an active infection.
* Pregnant (positive pregnancy test) or nursing women.
* Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy.
* Patients who have any disease that will obscure toxicity.
* Patients with evidence of acute intracranial/intratumoral hemorrhage on pre-study CT scan.
* Concurrent anti-coagulation or anti-platelet medication (including aspirin, -non-steroidal anti-inflammatories,
* cyclooxygenase 2 (COX-2) inhibitors).
* Serious or non-healing wound,
* ulcer
* or bone fracture
* History of abdominal fistula,
* gastrointestinal perforation
* or intra-abdominal abscess within 28 days
* Invasive procedures defined as follows:
* Major surgical procedure,
* open biopsy
* or significant traumatic injury within 28 days prior to Day 1 therapy
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to day 1 (D1) therapy
* Patients with clinically significant cardiovascular disease
* History of cerebrovascular accident (CVA) within 6 months
* Uncontrolled hypertension (greater than 150/100 mmHg)
* Myocardial infarction or unstable angina within 6 months
* New York Heart Association grade II or greater congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Unstable angina pectoris
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Prothrombin time (PT) international normalized ratio (INR) greater than 1.5
* Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-12; Primary Completion 2011-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teri Kreisl, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker D, Wright E, Nguyen K, Cannon L, Fain P, Goldgar D, Bishop DT, Carey J, Baty B, Kivlin J, et al. Gene for von Recklinghausen neurofibromatosis is in the pericentromeric region of chromosome 17. Science. 1987 May 29;236(4805):1100-2. doi: 10.1126/science.3107130.
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991
- [Result] Kreisl TN, Zhang W, Odia Y, Shih JH, Butman JA, Hammoud D, Iwamoto FM, Sul J, Fine HA. A phase II trial of single-agent bevacizumab in patients with recurrent anaplastic glioma. Neuro Oncol. 2011 Oct;13(10):1143-50. doi: 10.1093/neuonc/nor091. Epub 2011 Aug 24. PMID 21865400
- [Derived] Odia Y, Shih JH, Kreisl TN, Fine HA. Bevacizumab-related toxicities in the National Cancer Institute malignant glioma trial cohort. J Neurooncol. 2014 Nov;120(2):431-40. doi: 10.1007/s11060-014-1571-6. Epub 2014 Aug 7. PMID 25098701
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0064.html
- See also: Common Terminology Criteria for Adverse Events (CTCAE)v3.0 — http://ctep.cancer.gov
- See also: Response criteria for malignant gliomas — http://www.ncbi.nlm.nih.gov/pubmed/2358840
- See also: Criteria for malignant brain tumors — http://www.ncbi.nlm.nih.gov/pubmed/894339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 participants were accrued to this study.
Pre-assignment Details: Minimum washout period of 2-4 weeks required after molecularly targeted or cytotoxic agents.
Groups:
- Glioblastoma Multiforme (GBM): Glioblastoma multiforme Gliosarcoma
- Anaplastic Glioma (AG): Anaplastic astrocytoma Anaplastic oligodendroglioma Anaplastic mixed oligoastrocytoma Malignant astrocytoma (not otherwise specified)
Period: Overall Study
Arm/Group | Glioblastoma Multiforme (GBM) | Anaplastic Glioma (AG)
Started | 56 | 32
Completed | 43 | 29
Not Completed | 13 | 3
Not completed — Adverse Event | 11 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaplastic Glioma (AG) | Glioblastoma Multiforme (GBM) | Total
Number analyzed (Participants) | 32 | 56 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 50 | 80
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 52.33 (10.6) | 48.66 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 26 | 36
  Male | 22 | 30 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 29 | 55 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 28 | 55 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 56 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival at 6 Months.
Description: Percentage of participants surviving without progression of disease after six months of study entry. Progression is defined as a 25% increase in lesions, clear worsening of any evaluable disease, or appearance of any new lesion/site (e.g. by computed tomography, magnetic resonance imaging), or failure to return for evaluation due to death or deteriorating condition.
Time Frame: 6 months
Population: at the time of data cutoff for this endpoint, 31 patients in the AG arm and 48 patients in the GBM arm were evaluable for PFS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Anaplastic Glioma (AG) | Glioblastoma Multiforme (GBM)
Number analyzed (Participants) | 31 | 48
Percentage of participants | 20.9 [10.3 to 42.5] | 29 [18 to 48]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 5 years
Measure: Number; unit: Participants
Arm/Group | Anaplastic Glioma (AG) | Glioblastoma Multiforme (GBM)
Number analyzed (Participants) | 32 | 56
Participants | 32 | 51

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Anaplastic Glioma (AG) | Glioblastoma Multiforme (GBM)
Serious Adverse Events (participants affected / at risk) | 11/32 | 24/56
Other Adverse Events (participants affected / at risk) | 32/32 | 51/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Glioma (AG) (N=32) | Glioblastoma Multiforme (GBM) (N=56)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 7 (7)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 2 (2)
Death not associated with CTCAE term: death NOS (General disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term: disease progression NOS (General disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term: sudden death (General disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infection with normal ANC Grade 1 or 2 neutrophils: joint (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC: skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Investigations) | 0 (0) | 1 (2)
Lymphopenia (Investigations) | 0 (0) | 1 (1)
Musculoskeletal/soft tissue-other (specify-injury to the first index fingers & nail bed) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Necrosis, GI:gallbladder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 1 (1)
Opportunistic infection associated with >=Grade 2 lymphopenia (Infections and infestations) | 0 (0) | 2 (2)
Pain:headache (Nervous system disorders) | 0 (0) | 1 (2)
Pain:muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain:neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Perforation, GI: small bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils (Infections and infestations) | 1 (2) | 0 (0) — (ANC<1.0x10e9/L): Lung (pneumonia)
Infection with normal ANC or Grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Glioma (AG) (N=32) | Glioblastoma Multiforme (GBM) (N=56)
Hypertension (Vascular disorders) | 9 (12) | 11 (12)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 11 (15) | 11 (13)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 5 (6)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 11 (14) | 18 (28)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (6) | 10 (13)
Alkaline phosphatase (Investigations) | 1 (1) | 6 (7)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (2) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 1 (4) | 2 (2)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 9 (12) | 16 (32)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constitutional symptoms-other (Specify-orthostasis, "dizzines" when standing x minutes, self limited (General disorders) | 1 (1) | 0 (0)
Creatinine (Renal and urinary disorders) | 1 (9) | 1 (2)
Cushingoid appearance (e.g. moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Edema: limb (General disorders) | 3 (4) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Extremity-lower (gait/walking) (General disorders) | 1 (1) | 1 (1)
Gastrointestinal-Other (Specify-new urgency of bowel and bladder habits) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 6 (9) | 10 (14)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Rectum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L (Infections and infestations) | 1 (3) | 0 (0) — oral cavity-gums (gingivitis)
Infection with normal ANC or Grade 1 or 2 neutrophils: lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC Grade 1 or 2 neutrophils: nerve-peripheral (Infections and infestations) | 1 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: pharynx (Infections and infestations) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: sinus (Infections and infestations) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: skin (cellulitis) (Infections and infestations) | 2 (2) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: upper aerodigestive NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: upper airway NOS (Infections and infestations) | 4 (4) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils: urinary tract NOS (Infections and infestations) | 4 (7) | 2 (3)
Infection with unknown ANC: colon (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC: pharynx (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Lymphopenia (Investigations) | 8 (19) | 21 (49)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 7 (8) | 17 (26)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4) | 3 (6)
Memory impairment (Nervous system disorders) | 4 (4) | 1 (1)
Mood alteration: depression (Psychiatric disorders) | 5 (5) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)L extremity-lower (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 0 (0)
PTT (Partial thromboplastin Time) (Investigations) | 1 (2) | 5 (5)
Pain Other (Specify-pain-extremity-limb) (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain: Head/headache (Nervous system disorders) | 15 (25) | 11 (13)
Pain: joint (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5)
Pain: muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain: Neuralgia/peripheral nerve (Nervous system disorders) | 1 (1) | 0 (0)
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Pancreatic endocrine: glucose intolerance (Investigations) | 1 (2) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (16) | 19 (43)
Platelets (Investigations) | 10 (22) | 17 (29)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (7) | 3 (4)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 10 (27) | 24 (36)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1) | 2 (2)
Pulmonary/upper respiratory-Other (Specify-mild dry nasal mucosa) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyramidal tract dysfunction (Nervous system disorders) | 10 (12) | 5 (6) — (e.g. increased tone, hyperreflexia, positive Babinski, decreased fine coordination)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash: Hand/foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 1 (1)
Seizure (Vascular disorders) | 5 (5) | 13 (20)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 (15) | 10 (17)
Speech impairment (e.g. dysphasia or aphasia) (Nervous system disorders) | 4 (4) | 1 (1)
Supraventricular and nodal arrhythmia: sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (12) | 3 (6)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 2 (2)
Weight gain (Investigations) | 1 (1) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatology/Skin-Other (Specify-psoriasis) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (clinical exam): oral cavity (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neuropathy: Cranial-CN II vision (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 0 (0) | 1 (1)
Dermatology/skin-Other (Specify-tinea, requiring med. intervention) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eyelid dysfunction (Eye disorders) | 0 (0) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 5 (5)
Mucositis/stomatitis (functional/symptomatic): anus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neurology-Other (Specify-visual field cut) (Nervous system disorders) | 0 (0) | 1 (1)
Neurology: motor (Nervous system disorders) | 0 (0) | 1 (1)
Pain: Other (General disorders) | 0 (0) | 1 (1) — (Specify-during visit patient bent over to pick something up and had pain in L side in the lower rib area)
Pain: Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain : Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Prolonged QTc Interval (Cardiac disorders) | 0 (0) | 2 (2)
Rash: erythema multiforme (e.g. Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia: atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1)
Voice changes/dysarthria (e.g. hoarseness, loss or alteration in voice, laryngitis) (Vascular disorders) | 0 (0) | 4 (4)
Neurology-Other (Specify-worsening L-sided Parethesia, now clumsiness/?BCNU-related) (Nervous system disorders) | 1 (1) | 0 (0)
Rigors/Chills (General disorders) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: wound (Infections and infestations) | 0 (0) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils: Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (2)
Leukocytes (total WBC) (Investigations) | 0 (0) | 8 (13)
Fever ( in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1) | 0 (0)
Pain: oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Bicarbonate, serum low (Investigations) | 0 (0) | 3 (3)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemorrhage, GU: urinary NOS (Renal and urinary disorders) | 0 (0) | 4 (8)
Infection-Other (Specify- fungal infection with normal ANC) (Infections and infestations) | 0 (0) | 4 (4) — UTI (urinary tract infection) Whitish exudate on his tongue appeared to be thrush
Infection with unknown ANC: Upper airway NOS (Infections and infestations) | 1 (1) | 2 (2)
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1)
Mood alteration: Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy): extreme-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy): left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy): right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 3 (6)
Pain: neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC<1.0x10e9/L): mucosa
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage, Central nervous system (CNS) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Neuropathy-motor (Nervous system disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No